CLINICAL TRIAL: NCT03505684
Title: Effect of Oral Collagen Tripeptide on Skin Moisture and Wrinkles in Adult Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Sang Yeoup Lee, Principal Investigator, Professor, Head of Integrated Research Institute for Natural Ingredients and Functional Foods (IRINIF), Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 02-2017-033
Record Dates: First submitted 2018-04-13; First posted 2018-04-23 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Skin Manifestations; Skin Wrinkling
MeSH Terms: conditions — Skin Manifestations | interventions — Cytidine Triphosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTP group (Experimental): 1,000 mg of collagen tripeptide (CTP) was orally administered per day for 12 weeks.
  Interventions: Dietary Supplement: CTP
- Control group (Placebo Comparator): 1,000 mg of placebo (starch) was orally administered per day for 12 weeks
  Interventions: Dietary Supplement: placebo (starch)

INTERVENTIONS:
Dietary Supplement: CTP — 1,000 mg of CTP was orally administered per day for 12 weeks.
  Arms: CTP group
Dietary Supplement: placebo (starch) — placebo (starch)
  Arms: Control group

SUMMARY:
Comparison of a randomized, double-blind, and control-group study for the effect of oral ingestion of collagen tripeptides derived from fish on dermal moistures and wrinkles body fat reduction in participants

DETAILED DESCRIPTION:
The aim is to investigate the effect of oral ingestion of collagen tripeptides derived from fish on dermal moistures and wrinkles body fat reduction in participants by a randomized, double-blind, and control-group study.

ELIGIBILITY:
Inclusion Criteria:

- > = 4 of Tewameter

Exclusion Criteria:

* Within the last 6 months, took skin surgery including cosmetic purpose
* Diabetic patients with poor glycemic control with a fasting blood glucose of 160 mg/dl or more
* Creatinine levels: more than twice the normal upper limit
* AST (GOT) or ALT (GPT) levels: more than twice the normal upper limit
* Uncontrolled hypertension
* sun allergy or sensitive skin
* functional cosmetics that affect dermal moistures and wrinkles within the last 3 months.
* If you have participated or are planning to participate in another clinical trial within the past month
* Alcohol abuser
* If they are pregnant or lactating or have a pregnancy plan during the clinical trial Those with allergic reactions to the constituent food
* Any person deemed inappropriate by the researcher for other reasons

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2017-12-24 (Actual); Primary Completion 2018-07-15 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
changes in Transepidermal Waterloss by Tewameter | baseline, after 6 weeks, and after 12 weeks
  comparison between baseline, after 6 weeks, and after 12 weeks

SECONDARY OUTCOMES:
changes in skin wrinkling indices by Visiometer | baseline, after 6 weeks, and after 12 weeks
  comparison between baseline, after 6 weeks, and after 12 weeks
skin elasticity by Cutometer | baseline, after 6 weeks, and after 12 weeks
  comparison between baseline, after 6 weeks, and after 12 weeks
changes in hydration level of the skin surface by Corneometer | baseline, after 6 weeks, and after 12 weeks
  comparison between baseline, after 6 weeks, and after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sang Yeoup Lee, MD, Principal Investigator — Integrated Research Institute for Natural Ingredients and Functional Foods
Locations (1):
- Integrated Research Institute for Natural Ingredients and Functional Foods, Yangsan, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tak YJ, Shin DK, Kim AH, Kim JI, Lee YL, Ko HC, Kim YW, Lee SY. Effect of Collagen Tripeptide and Adjusting for Climate Change on Skin Hydration in Middle-Aged Women: A Randomized, Double-Blind, Placebo-Controlled Trial. Front Med (Lausanne). 2021 Jan 11;7:608903. doi: 10.3389/fmed.2020.608903. eCollection 2020. PMID 33521019